CLINICAL TRIAL: NCT00797264
Title: Impact of the Route of Administration of Ketamine Associated With Morphine PCA on Analgesia After Total Hip Arthroplasty
Brief Title: Ketamine Associated With Morphine PCA After Total Hip Arthroplasty
Acronym: KETAMINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P060402
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Ketamine; Morphine; PCA; Hyperalgesia; Nor-ketamine
MeSH Terms: conditions — Hyperalgesia | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Ketamine pre and per operative, and morphine postoperative
  Interventions: Drug: Ketamine-Morphine
- B (Active Comparator): NaCl pre and per operative, and morphine postoperative
  Interventions: Drug: Morphine
- C (Experimental): Ketamine and morphine postoperative
  Interventions: Drug: Postoperative PCA of Ketamine and morphine

INTERVENTIONS:
Drug: Ketamine-Morphine — Ketamine bolus preoperative and syringe pump peroperative, and morphine postoperative (PCA)
  Other Names: Ketamine pre and per operative, and morphine postoperative
  Arms: A
Drug: Morphine — Bolus preoperative of NaCl and syringe pump peroperative of NaCl, and morphine postoperative (PCA)
  Arms: B
Drug: Postoperative PCA of Ketamine and morphine — Bolus preoperative of NaCl and syringe pump peroperative of Ketamine, and morphine postoperative (PCA)
  Other Names: Ketamine Morphine
  Arms: C

SUMMARY:
Ketamine (an analgesic drug often associated with morphine in the treatment of Opioid Induced Hyperalgesia) is often mixed in Morphine PCA syringe. We make the hypothesis that ketamine administrated separately via a continuous infusion, could induced a better analgesic effect.

We will perform a randomised double blind study to determine the best infusion mode of intravenous ketamine, associated with morphine in PCA syringe or alone in continuous infusion.

DETAILED DESCRIPTION:
Double blind study to determine the best infusion mode of intravenous ketamine, associated with morphine in PCA syringe or alone in continuous infusion

ELIGIBILITY:
Inclusion Criteria:

* total hip arthroplasty

Exclusion Criteria:

* pre operative opioid administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Morphine consumption in PACU and in hospitalisation room | at 24 and 48 hours

SECONDARY OUTCOMES:
Postoperative Visual Analogic Score of pain | in Recovery Room, at 24 and 48 hours, in the ward
Postoperative Measure of mechanical hyperalgesia by Von Frey filament device | 24 and 48 hours in the ward
Postoperative measure Ketamine and Nor-Ketamine blood levels | at 24 and 48 hours in the ward

CONTACTS AND LOCATIONS:
Overall Officials: Philippe SITBON, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris Hôpital Bicêtre
Locations (1):
- Service d'anesthesie-reanimation - Hôpital Bicêtre, Le Kremlin-Bicêtre, France